CLINICAL TRIAL: NCT01633606
Title: Drawing the Line Between Medium Care and Intensive Care. A Prospective Observational Study Based on the Nursing Activities Score
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Greet Van den Berghe, professor, KU Leuven
Other Study IDs: NAS-ICU-2012
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Critical Illness
Keywords: severity of illness; scoring; medium care; intensive care; staffing
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute patients: Patients admitted to the surgical and general ICU (including burn unit), to the coronary care unit, to the emergency department high care zone, to the medical ICU, to the medical medium care unit

SUMMARY:
The aim of the study is to develop a screening instrument, based on the nursing activities score, by which we can distinguish medium care patients from the intensive care patients in terms of nurse staffing.

The main study question is: What is the most discriminative NAS cut off for medium care patient?

Each nursing shift the NAS and TISS 28 scores will be calculated for each patient who is admitted to the 8 participating units.

Nurses will be asked to answer 3 questions (see detailed description here under)at the end of their working shift concerning each patient appointed to them.

Each morning medical staff and head nurses will be asked 2 questions (see detailed description here under) for concerning patient admitted to there ward.

In order to determine the NAS cut off for medium care patient, all morning questionnaire scores will be compared to the NAS an TISS28 scores of that same morning.

Secondary study questions are:

* Can NAS score based on one nursing shift predict the severity of care in the subsequent nursing shift?
* Is there a difference in appreciation of severity of care between nurses, head nurses and medical staff?
* Which variables influence the perception of severity of care?
* How does NAS relate to TISS28, APACHE and NEMS?

DETAILED DESCRIPTION:
Nursing questionnaire:

1. How many beds were appointed to you?

   1. 1
   2. 2
   3. 3
   4. 4
   5. 5
   6. 6
2. For how many of such patients you could care for maximally?

   1. 1
   2. 2
   3. 3
   4. 4
   5. >4
3. This patients' burden of care corresponds to:

   1. An intensive care patient who requires more than standard intensive care
   2. An intensive care patient who requires standard intensive care
   3. A medium care patient

medical staff and head nurse questionaire:

1. For how many of such patients you could care for maximally?

   1. 1
   2. 2
   3. 3
   4. 4
   5. >4
2. This patients' burden of care corresponds to?

   1. An intensive care patient who requires more than standard intensive care
   2. An intensive care patient who requires standard intensive care
   3. A medium care patient

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the 9 critical area's

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
most discriminative NAS cut off for identifying medium care patient versus intensive care patient | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Greet Van den Berghe, MD PhD, Study Director — Catholic University Leuven; Karen Decock, RS, Principal Investigator — Universitaire Ziekenhuizen KU Leuven